CLINICAL TRIAL: NCT06629493
Title: Feasibility and Effects of Activity Trackers Among Alcohol Users Receiving In-patient Treatment for Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Alba González-Roz, PhD, Professor, PhD, University of Oviedo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SV-PA-21-AYUD/2021/50884(2)
Record Dates: First submitted 2024-07-30; First posted 2024-10-08 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2024-10

CONDITIONS: Substance-Related Disorders; Alcohol-Related Disorders; Alcohol Use Disorder (AUD)
Keywords: activity tracker; alcohol use disorder; physical activity; treatment; mental health
MeSH Terms: conditions — Substance-Related Disorders; Alcohol-Related Disorders; Alcoholism; Motor Activity; Psychological Well-Being | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alcohol use disorder treatment plus Fitbit Versa 3 (Experimental): Participants will receive in-patient treatment for alcohol use disorder plus an activity tracker
  Interventions: Behavioral: Fitbit Versa 3; Behavioral: In-patient alcohol use disorder treatment
- Alcohol use disorder treatment (Active Comparator): Participants will receive in-patient treatment for alcohol use disorder
  Interventions: Behavioral: In-patient alcohol use disorder treatment

INTERVENTIONS:
Behavioral: Fitbit Versa 3 — Fitbit Versa 3 is a commercially available activity tracker
  Arms: Alcohol use disorder treatment plus Fitbit Versa 3
Behavioral: In-patient alcohol use disorder treatment — In-patient alcohol use disorder treatment, including group therapy, counseling, and occupational activities

SUMMARY:
The main objective is to assess the feasibility and effectiveness of using activity trackers to increase physical activity and improve the emotional state of people receiving an in-patient treatment for alcohol use disorder

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years old or older.
* Be undergoing inpatient treatment for alcohol use disorder.

Exclusion Criteria:

* Finishing the treatment before 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Physical activity tracker adherence | Treatment duration (4 weeks)
  Days (percentage) in which activity tracker was used (day-time and night-time use)
Physical activity tracker perceived utility | End-of-treatment (4 weeks)
  Perceived utility with the physical activity tracker will be assessed using ad-hoc questions about the utility of the activity tracker to increase levels of physical activity, improve sleep quality, and reduce/abandon tobacco.
Physical activity levels | In-treatment (4 weeks), from enrollment to end-of treatment (4 weeks)
  Physical activity (PA) is operationalized as steps per day, plants climbed per day, distance covered per day (kilometers), light physical activity (minutes per day), moderate physical activity (minutes per week), vigorous physical activity (minutes per week), and sedentary time (hours per day). These outcomes will be measured using an adapted version of the International Physical Activity Questionnaire (IPAQ) and Fitbit Versa 3®.
Depression symptoms | From enrollment to the end-of-treatment (4 weeks)
  Depression symptoms will be measured using the Patient Health Questionnaire-9 (PHQ-9). This questionnaire ranges from 0 to 14. A higher punctuation means higher depression symptom levels.
Anxiety symptoms | From enrollment to the end-of-treatment (4 weeks)
  Anxiety symptoms will be measured using Generalized Anxiety Disorder-7 (GAD-7). This questionnaire ranges from 0 to 21. Higher punctuation means higher anxiety levels symptoms.
Difficulties in emotion regulation | From enrollment to the end-of-treatment (4 weeks)
  Emotion dysregulation is measured using the Difficulties in Emotion Regulation Scale (DERS). Emotional dysregulation of negative emotions is measured with the Difficulties in Emotion Regulation Scale (DERS). This scale ranges from 28 to 140 points. A higher score means more difficulties in emotion regulation.
Physical activity tracker acceptability | End-of-treatment (4 weeks)
  Acceptability of the activity tracker is measured using the Participant Experience Questionnaire (PEQ). This scale ranges from 10 to 50 points. A higher score means higher acceptability.
Sleep quality | In-treatment (4 weeks), from enrollment to the end-of-treatment (4 weeks)
  Sleep quality will be measured using both the Pittsburg Sleep Quality Index (PSQI) and the Fitbit Versa 3. PSQI ranges from 0 to 21 points. A higher score means lower sleep quality. In addition, Fitbit Versa 3 provides a sleep quality punctuation ranging from 0 to 100. A higher punctuation means better sleep quality.

SECONDARY OUTCOMES:
Tobacco use | In treatment (4 weeks), from enrollment to the end-of-treatment (4 weeks)
  Self-reported cigarettes per day and carbon monoxide (CO) levels measured by a CO monitor reading.
Delay discounting (impulsive decision making) | From enrollment to the end-of-treatment (4 weeks)
  Delay discounting will be measured using the 21-item Monetary-Choice task. Computerized Delay Discounting task of tobacco (delay of one day, one week, one month, and six months).

CONTACTS AND LOCATIONS:
Locations (1):
- Therapeutical community "La Santina", Gijón, Principality of Asturias, Spain

REFERENCES:
- [Background] Scott CK, Dennis ML, Gustafson DH. Reprint of Using ecological momentary assessments to predict relapse after adult substance use treatment. Addict Behav. 2018 Aug;83:116-122. doi: 10.1016/j.addbeh.2018.04.003. Epub 2018 Apr 7. PMID 29661655
- [Background] Purani H, Friedrichsen S, Allen AM. Sleep quality in cigarette smokers: Associations with smoking-related outcomes and exercise. Addict Behav. 2019 Mar;90:71-76. doi: 10.1016/j.addbeh.2018.10.023. Epub 2018 Oct 17. PMID 30368021
- [Background] Brickwood KJ, Watson G, O'Brien J, Williams AD. Consumer-Based Wearable Activity Trackers Increase Physical Activity Participation: Systematic Review and Meta-Analysis. JMIR Mhealth Uhealth. 2019 Apr 12;7(4):e11819. doi: 10.2196/11819. PMID 30977740
- [Background] Abrantes AM, Blevins CE, Battle CL, Read JP, Gordon AL, Stein MD. Developing a Fitbit-supported lifestyle physical activity intervention for depressed alcohol dependent women. J Subst Abuse Treat. 2017 Sep;80:88-97. doi: 10.1016/j.jsat.2017.07.006. Epub 2017 Jul 8. PMID 28755778
- See also: Fitbit webpage, where information about the the device used in the trial can be found — https://www.fitbit.com/global/es/home